CLINICAL TRIAL: NCT06899503
Title: CLICK: Creating Linked Inpatient CGM for Kids
Brief Title: Creating Linked Inpatient CGM for Kids
Acronym: CLICK
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jessica Ruiz, MD, Physician, Endocrinology, Boston Children's Hospital
Other Study IDs: IRB-P00049941
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Diabetes; Continuous Glucose Monitoring System
Keywords: Diabetes; Continuous glucose monitoring system; Android application
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric diabetic Dexcom G7 users: Diabetic pediatric patients using their personal Dexcom G7 admitted for clinical care purposes.

SUMMARY:
Continuous glucose monitors (CGMs) are currently used in the inpatient setting at many hospitals for the care of patients with diabetes and for clinical research studies. This includes Boston Children's Hospital, however, the CGM data is not accessible to clinical or research teams in real-time. CGMs measure and display a patient's glucose level every 5 minutes and provide alerts for predicted or actual low or high glucose levels. The CGM data is currently only accessible on bedside handheld receivers or a mobile device app, neither of which sync with the hospital EMR or other hospital databases. This observational study tests a companion mobile Android device app that wirelessly receives real-time outputs from the Dexcom G7 CGM app and transmits the data to a centralized hospital database. That database in turn feeds into an internal BCH web dashboard which allows live data viewing and integration into future clinical decision support tools.

The investigators are testing the hypothesis that the companion mobile app can accurately and efficiently transmit CGM data to a hospital database. Data will be analyzed for accuracy and efficiency by comparing CGM readings captured by the companion app to CGM readings documented in the formal Dexcom database. Accuracy (difference between CGM readings from both sources) and efficiency (number of CGM readings captured) will be assessed. The findings will be generalizable to using the companion app in future research studies.

DETAILED DESCRIPTION:
Continuous glucose monitors are currently used in the inpatient setting at Boston Children's Hospital (BCH) for the care of patients with diabetes and for research studies. CGMs measure and display patient's glucose level every 5 minutes and provide alerts for predicted or actual low or high glucose levels. BCH policy allows for use of Dexcom G6 and G7 CGM for glucose monitoring and insulin dosing, so long as the CGM accuracy is verified daily.

Currently, CGM data is not accessible to clinical or research teams in real-time. The CGM data is currently only accessible on bedside handheld receivers or a cell phone app, neither of which syncs with the hospital EMR or other hospital databases. The current clinical workflow requires the bedside caregiver to alert the clinical team of any glucose abnormalities. In order to view and document CGM glucose levels in real-time, clinical and research teams must be physically at the bedside viewing the CGM receiver or the patient's personal cell phone app screen. Teams do have access to the Dexcom Clarity database, an online cloud-based data viewing dashboard, but data transmission is delayed 3 hours from the Dexcom cloud database to Dexcom Clarity.

This observational study tests a companion mobile Android application that receives real-time data from the Dexcom G7 CGM app running on a hospital provided mobile device. The companion app and G7 app modifications were developed from a protocol created by patients in the diabetes community who wanted expanded access to their own data, and was adapted by BCH co-investigators to work entirely within the BCH firewall to access and share the data within BCH. Investigators will recruit individuals using their personal Dexcom G7 CGM in the hospital for clinical care, have the participants use the Dexcom G7 app on a hospital provided Android device, and will test the accuracy and efficiency of data capture by the companion app, all via secure BCH wifi or ethernet. On the hospital device, the Dexcom G7 app has been modified to send Android intra-application messages with CGM readings without identifying information to a companion app. The companion app will transmit the de-identified CGM data to a centralized hospital database that feeds into an internal BCH web dashboard for live data viewing, analysis, and integration into future clinical decision support tools. One anticipated future use of the companion app will be in an upcoming interventional clinical trial of ICU patients receiving IV insulin, in which CGM data will be used to guide insulin infusion rates.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with diabetes using a Dexcom G7 CGM
* Technology/data sharing criteria: use of the Dexcom G7 phone app and data sharing with the BCH Dexcom Clarity Database
* Anticipated discharge date >24 hours after study eligibility

Exclusion Criteria:

* Use of medications that interfere with CGM accuracy
* Use of a Dexcom receiver to view data (rather than the typical mobile phone)
* Enrollment in a competing clinical trial

Ages: 2 Weeks to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inpatients at Boston Children's Hospital (BCH) with diabetes, admitted for clinical care purposes, using their personal Dexcom G7 CGM during the inpatient admission.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of CGM data capture. | The earlier of a maximum of 20 days or 72 hours following the first sensor exchange.
  The accuracy of the CGM readings captured will be measured as the mean absolute relative difference (MARD) between the CGM glucose reading captured by the companion app compared to the CGM glucose reading documented in the Dexcom Clarity database within the same 5-minute interval.

SECONDARY OUTCOMES:
Efficiency of CGM data capture. | The earlier of a maximum of 20 days or 72 hours following the first sensor exchange.
  Efficiency of CGM data capture, measured as the percent of CGM readings documented in Dexcom Clarity that were also captured by the companion app within the same 5-minute interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No